CLINICAL TRIAL: NCT04843956
Title: Comparación de Tres técnicas de Biopsia Guiada Por Endosonografia de Lesiones sólidas pancreáticas
Brief Title: Comparison of EUS-FNB Biopsy Techniques of Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical profesor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GA19-00014
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Masking Description: The samples will be analyzed independently by the pathology service, not knowing the order and the technique in which the samples were obtained. The histopathological result will be immediately available for patient care, however, the score obtained regarding the quality of the sample will correlate with the technique and the number of passes until the n of the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with solid pancreatic lesions (Experimental): Patients who will undergo endoscopic ultrasound biopsy. Samples of at least 3 passes will be obtained, each pass obtained with a different technique (capillary with suction, capillary without suction and wet suction)
  Interventions: Diagnostic Test: Endoscopic ultrasound-guided biopsy

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound-guided biopsy — Capillary with suction (puncture with gradual withdrawal of the stylet, applying dry suction with a 10 ml air vacuum syringe after removing the stylet)
  Capillary without suction (puncture with removal of the stylet gradually, without suction after removing the stylet)
  wet suction (Prior to puncture, the stylet is removed from the needle and irrigated with 1-2 ml saline solution to replace the air column with liquid, then the solid lesion is punctured and suction is placed with a 10 ml vacuum syringe of air)
  Other Names: Pancreatic biopsy

SUMMARY:
Patients with a diagnosis of solid pancreatic lesions evidenced by imaging studies (CT, MRI) and who undergo endoscopic ultrasound-guided biopsy will be selected. Biopsies will be taken using modified tip needles (FNB) three different methods (capillary by suction, capillary without suction and wet suction).

From the results obtained from the pathology service, 3 variables will be assessed; Cellularity, blood contamination and suitability for a diagnosis.

DETAILED DESCRIPTION:
EUS-BAAF procedure The procedure will be performed with a linear echoendoscope (PENTAX 3.8 EG-3870 UTK) and a HITACHI HI VISION Avius ultrasound processor, after deep sedation by the anesthesiology service. BAF Acquire # 22 needles (Boston Scientific, Malborough, MA) will be used. 3 passes will be made to the tumor, each pass will consist of 10-15 movements of the needle back and forth in a fan within the solid lesion, under complete ultrasound control (ESGE 2017- Gastrointest Endoscopy Clin N Am 22 (2012) 155 -167). Doppler will be used to avoid any vascular structure in the path of the needle.

The passes will be in three different ways to compare.

1. Capillary with suction (puncture with gradual withdrawal of the stylet, applying dry suction with a 10 ml air vacuum syringe after removing the stylet)
2. Capillary without suction (puncture with removal of the stylet gradually, without suction after removing the stylet)
3. Moist suction (Before the puncture, the stylet is removed from the needle and irrigated with 1-2 ml saline solution to replace the air column with liquid, then the solid lesion is punctured and suction is placed with a vacuum syringe of 10 ml of air)

The quality of the biopsy will be evaluated by the pathologist independently and without knowing how the sample was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Any gender.
* Patients with solid pancreatic lesions evidenced by CT or MRI who do not have a histopathological diagnosis.

Exclusion Criteria:

* That no lesion in the pancreas is identified by EUS.
* Pancreatic lesions with a cystic component.
* Alteration of coagulation parameters (INR> 1.5, Platelets <50,000 / mm3) or having taken antiplatelet agents or oral anticoagulants one week prior to the biopsy.
* History of acute pancreatitis in the last 4 weeks.
* Pregnant
* Refusal or inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of the sample in relation to the technique | 18 months
  Establish if there is a difference in the quality of the sample in relation to the technique used to obtain it

SECONDARY OUTCOMES:
Sample contamination relative to technique | 18 months
  Establish if there is a difference in the contamination of the sample, in relation to the technique used to obtain it

CONTACTS AND LOCATIONS:
Locations (1):
- Héctor Miguel Delgado Cortes, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
No individual data sharing plan

REFERENCES:
- [Background] Lee YN, Moon JH, Kim HK, Choi HJ, Choi MH, Kim DC, Lee TH, Cha SW, Cho YD, Park SH. Core biopsy needle versus standard aspiration needle for endoscopic ultrasound-guided sampling of solid pancreatic masses: a randomized parallel-group study. Endoscopy. 2014 Dec;46(12):1056-62. doi: 10.1055/s-0034-1377558. Epub 2014 Aug 6. PMID 25098611
- [Background] Crino SF, Manfrin E, Scarpa A, Baldaque-Silva F, Carrara S, De Nucci G, Di Mitri R, Gines A, Iglesias-Garcia J, Itoi T, Kitano M, Nguyen NQ, Deprez PH, Poley JW, Shami VM, Tarantino I, Larghi A. EUS-FNB with or without on-site evaluation for the diagnosis of solid pancreatic lesions (FROSENOR): Protocol for a multicenter randomized non-inferiority trial. Dig Liver Dis. 2019 Jun;51(6):901-906. doi: 10.1016/j.dld.2019.03.008. Epub 2019 Apr 8. PMID 30975612
- [Background] Bor R, Vasas B, Fabian A, Balint A, Farkas K, Milassin A, Czako L, Rutka M, Molnar T, Szucs M, Tiszlavicz L, Kaizer L, Hamar S, Szepes Z. Prospective comparison of slow-pull and standard suction techniques of endoscopic ultrasound-guided fine needle aspiration in the diagnosis of solid pancreatic cancer. BMC Gastroenterol. 2019 Jan 9;19(1):6. doi: 10.1186/s12876-018-0921-9. PMID 30626331
- [Background] Aadam AA, Oh YS, Shidham VB, Khan A, Hunt B, Rao N, Zhang Y, Tarima S, Dua KS. Eliminating the Residual Negative Pressure in the Endoscopic Ultrasound Aspirating Needle Enhances Cytology Yield of Pancreas Masses. Dig Dis Sci. 2016 Mar;61(3):890-9. doi: 10.1007/s10620-015-3860-0. Epub 2015 Sep 7. PMID 26346997
- [Background] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878
- [Background] Kudo T, Kawakami H, Hayashi T, Yasuda I, Mukai T, Inoue H, Katanuma A, Kawakubo K, Ishiwatari H, Doi S, Yamada R, Maguchi H, Isayama H, Mitsuhashi T, Sakamoto N; Japan EUS-FNA Negative Pressure Suction Study Group. High and low negative pressure suction techniques in EUS-guided fine-needle tissue acquisition by using 25-gauge needles: a multicenter, prospective, randomized, controlled trial. Gastrointest Endosc. 2014 Dec;80(6):1030-7.e1. doi: 10.1016/j.gie.2014.04.012. Epub 2014 Jun 2. PMID 24890422
- [Background] Bansal RK, Choudhary NS, Puri R, Patle SK, Bhagat S, Nasa M, Bhasin A, Sarin H, Guleria M, Sud R. Comparison of endoscopic ultrasound-guided fine-needle aspiration by capillary action, suction, and no suction methods: a randomized blinded study. Endosc Int Open. 2017 Oct;5(10):E980-E984. doi: 10.1055/s-0043-116383. Epub 2017 Oct 4. PMID 28983505
- [Background] Li H, Li W, Zhou QY, Fan B. Fine needle biopsy is superior to fine needle aspiration in endoscopic ultrasound guided sampling of pancreatic masses: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Mar;97(13):e0207. doi: 10.1097/MD.0000000000010207. PMID 29595661
- [Background] Polkowski M, Jenssen C, Kaye P, Carrara S, Deprez P, Gines A, Fernandez-Esparrach G, Eisendrath P, Aithal GP, Arcidiacono P, Barthet M, Bastos P, Fornelli A, Napoleon B, Iglesias-Garcia J, Seicean A, Larghi A, Hassan C, van Hooft JE, Dumonceau JM. Technical aspects of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Guideline - March 2017. Endoscopy. 2017 Oct;49(10):989-1006. doi: 10.1055/s-0043-119219. Epub 2017 Sep 12. PMID 28898917
- [Background] Ge PS, Wani S, Watson RR, Sedarat A, Kim S, Marshall C, Wilson RH, Makker J, Mohamadnejad M, Komanduri S, Muthusamy VR. Per-Pass Performance Characteristics of Endoscopic Ultrasound-Guided Fine-Needle Aspiration of Malignant Solid Pancreatic Masses in a Large Multicenter Cohort. Pancreas. 2018 Mar;47(3):296-301. doi: 10.1097/MPA.0000000000001003. PMID 29401169